CLINICAL TRIAL: NCT02372734
Title: Long Term Cognitive Impact of Pediatric Acute Renal Injury
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Society of Nephrology (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401054
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis with acute kidney injury (AKI): Prior admission for sepsis with a diagnosis of AKI as a child. Intervention: The subjects will be administered the Peds QL survey.
  Interventions: Other: Pediatric Quality of Life (Peds QL) Survey
- Sepsis without acute kidney injury (AKI): Prior admission for sepsis without a diagnosis of AKI as a child. Intervention: The subjects will be administered the Peds QL survey.
  Interventions: Other: Pediatric Quality of Life (Peds QL) Survey

INTERVENTIONS:
Other: Pediatric Quality of Life (Peds QL) Survey — The subjects will be administered the Peds QL survey. Children will also have a parental section for parental response. This is NOT an interventional study.

SUMMARY:
The research study will investigate the longitudinal cognitive outcomes in subjects admitted as children diagnosed with sepsis who may have had acute kidney injury. Each subject will be contacted 2-15 years after their incident admission in order to solicit responses to a functional and cognitive quality of life survey. Children admitted during the same time frame that did not have kidney injury will also be surveyed.

DETAILED DESCRIPTION:
250 subjects with a prior admission for pediatric sepsis will be contacted 2-15 years following the incident admission in order to complete a survey to assess their overall quality of life. Children will be administered the Pediatric Quality of Life (PedsQL) survey with a parental section to allow for parental response. Adult subjects will take the adult version of the PedsQL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be adults or children who were admitted to the hospital with a severe infection between January 1998 to December 2014.
* Consent from adult or parent/guardian of child to participate in study.
* Assent from subjects between 7 and 17 years of age.

Exclusion Criteria:

* Failure or inability to complete the survey
* Participant is unable to understand written or spoken English
* Subjects between 7 and 17 years of age unwilling to assent.

Ages: 2 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects are former patients admitted for sepsis as a child.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Overall health related quality of life score (HRQOL) | Baseline
  Scale 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Carmelle Elie, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States